CLINICAL TRIAL: NCT03480581
Title: Impact of Reverse vs. Forward ICARE Training Interventions on Walking and Fitness of Individuals With Walking Disorders Arising From Neurologic Injuries or Illnesses
Brief Title: Impact of Reverse vs. Forward ICARE Training Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Madonna Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Judith M. Burnfield, PhD, PT, Director, Institute for Rehabilitation Science and Engineering, Madonna Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18-001-FB
Record Dates: First submitted 2018-03-07; First posted 2018-03-29 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Neurological Injury; Neurological Diseases or Conditions
Keywords: Neurological; Gait; Cardiorespiratory fitness; Rehabilitation; Walking; Locomotor training; Robotics
MeSH Terms: conditions — Trauma, Nervous System; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reverse First ICARE Training (Experimental): Participants will engage in 12-sessions in the reverse direction followed by 12-sessions in the forward direction.
  Interventions: Behavioral: Reverse First ICARE Training
- Forward First ICARE Training (Experimental): Participants will engage in 12-sessions in the forward direction followed by 12-sessions in the reverse direction.
  Interventions: Behavioral: Forward First ICARE Training

INTERVENTIONS:
Behavioral: Forward First ICARE Training — Participants will engage in 12-sessions in forward direction, followed by 12-sessions in the reverse direction. Sessions will be scheduled 3 times/week with training parameters adjusted to progressively increase challenge as tolerated.
  Arms: Forward First ICARE Training
Behavioral: Reverse First ICARE Training — Participants will engage in 12-sessions in reverse direction, followed by 12-sessions in the forward direction. Sessions will be scheduled 3 times/week with training parameters adjusted to progressively increase challenge as tolerated.
  Arms: Reverse First ICARE Training

SUMMARY:
The goal of this study is to determine if training in both the forward and reverse modes on the ICARE (motor-assisted elliptical) contributes to improvements in gait and cardiorespiratory fitness.

DETAILED DESCRIPTION:
A growing number of facilities are using the robotic ICARE, a motor-assisted elliptical, to improve walking and fitness in individuals with physical disabilities. The device promotes movements emulating the joint motions and muscle demands of normal gait and integrates design features that improve accessibility and usability (e.g., motor assistance, partial BWS, electronic height-adjustable seat, steps, ramp, wheelchair platform) compared to traditional ellipticals. A motor assists those with strength and/or endurance limitations to train (forward/reverse directions) at speeds up to 65 cycles per minute (CPM), thus creating opportunities for the mass repetition of a gait-like movement pattern that is often advocated as critical for behavioral and neurologic recovery. Individuals can over-ride the motor's assistance simply by training faster than the set speed. Documented improvements in walking and cardiorespiratory fitness in individuals with neurologic injuries and illnesses following an ICARE training program in the forward direction are promising.

Reverse walking is one method clinicians have used to improve forward walking performance in patients with various neurological disorders. Although the ICARE allows for reverse training, and this feature has been used clinically, no studies to date have compared changes in walking and cardiorespiratory fitness arising from an ICARE training intervention performed in the reverse direction to those arising from an ICARE intervention performed in the forward direction. Thus, the purpose of this exploratory study is to compare gait and cardiorespiratory improvements arising from blocks (12-sessions) of forward vs. reverse ICARE training in participants with walking dysfunction. For this exploratory study, the investigators hypothesize that both forward and reverse training will contribute to improvements in gait and cardiorespiratory fitness. In addition, the investigators seek to understand whether the magnitude of change will differ between each form of training (i.e., forward vs. reverse) and whether the order of training will impact the magnitude of change (i.e. block of 12-sessions forward followed by block of 12-sessions reverse vs. block of 12-sessions reverse followed by block of 12-sessions forward). Measurements will be recorded immediately prior to intervention initiation (T0), following completion of the first training block (T1), immediately following completion of the second training block (T2), and 3 months following completion of the second training block (T3)

ELIGIBILITY:
Inclusion Criteria:

* Walking dysfunction from a neurologic injury or illness (e.g. stroke, brain injury, incomplete spinal cord injury, multiple sclerosis, Parkinson's disease, cerebral palsy);
* Able to stand (with or without a standing frame) for at least 5 minutes at a time;
* Able to follow simple commands; and
* Possess adequate judgment or communication skills to safely use the ICARE trainer.

Exclusion Criteria:

* Currently enrolled in an existing physical or occupational therapy program or an exercise program for their legs;
* Orthopedic conditions (such as bone fractures/breaks) that haven't healed;
* Unstable cardiac or respiratory conditions that would prohibit safe exercise;
* Pregnant or think they may be pregnant, given unknown but potential risk of vigorous exercise to the mother and/or the unborn fetus; and/or
* Experience self-reported pain that inhibits walking/exercise ability.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
10 Meter Walk Test Speed | 10 minutes
  Average walking speed while traversing 10 meters
Peak Oxygen Consumption | Up to 30 minutes
  This test of aerobic capacity quantifies the peak oxygen consumed while walking on a treadmill or rotating a crank ergometer

SECONDARY OUTCOMES:
6 Minute Walk Test | Up to 2 minute explanation followed by 6 minute formal walk test
  This sub-maximal exercise test measures the maximum distance walked during 6 minutes. It is used to assess aerobic capacity and endurance. Protocol includes 2 minute explanation followed by 6 Minute Walk Test.
Energy Cost of Treadmill Walking | Up to 30 minutes
  This metabolic test of walking efficiency measures oxygen consumed during treadmill walking and divides it by the treadmill's walking speed.
Cardiorespiratory Response During Treadmill Walking | Up to 30 minutes
  Ratings of perceived effort during graded exercise test
Cardiorespiratory Response During ICARE Training | Up to 50 minutes
  Ratings of perceived effort while training on the ICARE
Spatiotemporal Gait Measures | 20 minutes
  Stride characteristics (e.g., cadence, stride length, single limb support time) recorded while traversing instrumented walkway
Timed Up and Go (TUG) Test | 8 minutes
  Time required to completed standardized TUG test, a measure used to assess a person's mobility that requires both static and dynamic balance.

CONTACTS AND LOCATIONS:
Overall Officials: Judith M. Burnfield, Ph.D., Principal Investigator — Madonna Rehabilitation Hospital
Locations (1):
- Madonna Rehabilitation Hospital, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan for sharing IPD.

REFERENCES:
- [Background] Burnfield JM, Shu Y, Buster TW, Taylor AP, Nelson CA. Impact of elliptical trainer ergonomic modifications on perceptions of safety, comfort, workout, and usability for people with physical disabilities and chronic conditions. Phys Ther. 2011 Nov;91(11):1604-17. doi: 10.2522/ptj.20100332. Epub 2011 Sep 1. PMID 21885449
- [Background] Burnfield JM, Shu Y, Buster T, Taylor A. Similarity of joint kinematics and muscle demands between elliptical training and walking: implications for practice. Phys Ther. 2010 Feb;90(2):289-305. doi: 10.2522/ptj.20090033. Epub 2009 Dec 18. PMID 20022994
- [Background] Burnfield JM, Cesar GM, Buster TW, Irons SL, Nelson CA. Kinematic and muscle demand similarities between motor-assisted elliptical training and walking: Implications for pediatric gait rehabilitation. Gait Posture. 2017 Jan;51:194-200. doi: 10.1016/j.gaitpost.2016.10.018. Epub 2016 Oct 24. PMID 27810692
- [Background] Burnfield JM, Irons SL, Buster TW, Taylor AP, Hildner GA, Shu Y. Comparative analysis of speed's impact on muscle demands during partial body weight support motor-assisted elliptical training. Gait Posture. 2014;39(1):314-20. doi: 10.1016/j.gaitpost.2013.07.120. Epub 2013 Aug 3. PMID 23973354
- [Background] Buster T, Burnfield J, Taylor AP, Stergiou N. Lower extremity kinematics during walking and elliptical training in individuals with and without traumatic brain injury. J Neurol Phys Ther. 2013 Dec;37(4):176-86. doi: 10.1097/NPT.0000000000000022. PMID 24189335
- [Background] Kim SG, Ryu YU, Je HD, Jeong JH, Kim HD. Backward walking treadmill therapy can improve walking ability in children with spastic cerebral palsy: a pilot study. Int J Rehabil Res. 2013 Sep;36(3):246-52. doi: 10.1097/MRR.0b013e32835dd620. PMID 23370765
- [Background] Yang YR, Yen JG, Wang RY, Yen LL, Lieu FK. Gait outcomes after additional backward walking training in patients with stroke: a randomized controlled trial. Clin Rehabil. 2005 May;19(3):264-73. doi: 10.1191/0269215505cr860oa. PMID 15859527
- [Background] Irons, S.L., et al., Novel motor-assisted elliptical training intervention improves Six-Minute Walk Test and oxygen cost for an individual with progressive supranuclear palsy. Cardiopulmonary Physical Therapy Journal, 2015. 26(2): p. 36-41.
- [Background] Nelson, C.A., et al., Modified elliptical machine motor-drive design for assistive gait rehabilitation. Journal of Medical Devices, 2011. 5(June): p. 021001.1-7.
- [Background] Nelson, C.A., et al., Modification of the Intelligently Controlled Assistive Rehabilitation Elliptical (ICARE) system for pediatric therapy. Published online, ASME Journal of Medical Devices. DOI: 10.1115/1.4030276., 2015.
- [Background] Irons, S.L., et al., Individuals with multiple sclerosis improved walking endurance and decreased fatigue following motor-assisted elliptical training intervention [Abstract]. Archives of Physical Medicine and Rehabilitation, 2016. 97(10): p. e34.
- [Background] Burnfield, J.M., et al., Pedi-ICARE training improves walking and endurance of child with cerebral palsy. Archives of Physical Medicine and Rehabilitation, 2016. 97(12): p. E19-E20.
- [Background] Cesar, G.M., et al., Child with traumatic brain injury improved gait abilities following intervention with pediatric motor-assisted elliptical training: A case report. Journal of Neurologic Physical Therapy, 2017. 41(1): p. 84.